CLINICAL TRIAL: NCT05029089
Title: Modified Entire Papilla Preservation Technique (MEPPT) For Periodontal Regenerative Treatment Of Intrabony Defects. A Randomized Clinical Trial.
Brief Title: Modified Entire Papilla Preservation Technique For Treatment Of Intrabony Defects. Clinical Trial.
Acronym: MEPPT
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Medical University of Warsaw (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: WUM.Perio.04
Record Dates: First submitted 2021-07-19; First posted 2021-08-31 (Actual); Last update posted 2021-10-12 (Actual); Status verified 2021-08

CONDITIONS: Periodontitis; Regeneration
Keywords: Papilla Preservation Technique; Regenerative Treatment; Allograft; Emdogain
MeSH Terms: conditions — Periodontitis | interventions — Transplantation, Homologous

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Experimental: Entire Papilla Preservation Modified Technique (EPPMT) (Experimental): Procedure: The surgical site was anesthetized with articaine-epinephrine. After buccal intracervicular incision on vestibular aspects of two teeth surrounding the intrabony defect, a beveled vertical releasing incision was made in the buccal gingiva of the tooth affected by the intrabony defect, on the opposite site to the intrabony defect and extended beyond the mucogingival line to provide access to the intrabony defect. A buccal full thickness mucoperiosteal flap extending from the vertical incision to the defect-associated papilla and neigboring tooth was elevated (subperiosteal tunnel). Interdental tunnel under the papillary tissue was elevated to the lingual bone crest. Granulation tissue and calculus from the inner aspect of interdental papilla was removed. Microsurgical suturing technique with 7-0 materials was performed. Vertical incision was closed with simple single sutures, whereas due to modification of the original technique additional sling suture was applied.
  Interventions: Procedure: Modified Entire Papilla Preservation Technique (MEPPT) For Periodontal Regenerative Treatment Of Intrabony Defects.
- Entire Papilla Preservation Modified Technique + EMD (Active Comparator): Procedure: The surgical site was anesthetized with articaine-epinephrine. After buccal intracervicular incision on vestibular aspects of two teeth surrounding the intrabony defect, a beveled vertical releasing incision was made in the buccal gingiva of the tooth affected by the intrabony defect, on the opposite site to the intrabony defect and extended beyond the mucogingival line to provide access to the intrabony defect. A buccal full thickness mucoperiosteal flap extending from the vertical incision to the defect-associated papilla and neigboring tooth was elevated. Interdental tunnel under the papillary tissue was elevated to the lingual bone crest. Granulation tissue and calculus from the inner aspect of interdental papilla was removed. 24%EDTA was applied on the exposed root surface for 2 minutes, than rinsed and EMD was applied. Vertical incision was closed with simple single sutures(7-0),whereas due to modification of the original technique additional sling suture was applied.
  Interventions: Procedure: Modified Entire Papilla Preservation Technique (MEPPT) For Periodontal Regenerative Treatment Of Intrabony Defects.; Device: Emdogain (EMD), Biomaterials (allograft, subepithelial connective tissue graft/sCTG); Procedure: Modified Entire Papilla Preservation Technique (MEPPT) with Emdogain For Periodontal Regenerative Treatment Of Intrabony Defect
- EPP Modified Technique+EMD+allograft (Active Comparator): Procedure:The surgical site was anesthetized with articaine-epinephrine. After buccal intracervicular incision on vestibular aspects of two teeth surrounding the intrabony defect, a beveled vertical releasing incision was made in the buccal gingiva of the tooth affected by the intrabony defect, on the opposite site to the intrabony defect and extended beyond the mucogingival line to provide access to the intrabony defect. A buccal full thickness mucoperiosteal flap extending from the vertical incision to the defect-associated papilla and neigboring tooth was elevated. Interdental tunnel under the papillary tissue was elevated to the lingual bone crest. Granulation tissue and calculus from the inner aspect of interdental papilla was removed.24%EDTA was applied on the exposed root surface, than rinsed and EMD and bone substitute was applied. Vertical incision was closed with simple single sutures, whereas due to modification of the original technique additional sling suture was applied.
  Interventions: Procedure: Modified Entire Papilla Preservation Technique (MEPPT) For Periodontal Regenerative Treatment Of Intrabony Defects.; Device: Emdogain (EMD), Biomaterials (allograft, subepithelial connective tissue graft/sCTG); Procedure: Modified Entire Papilla Preservation Technique (MEPPT) with Emdogain For Periodontal Regenerative Treatment Of Intrabony Defect; Procedure: Modified Entire Papilla Preservation Technique (MEPPT) with Emdogain and Allograft For Periodontal Regenerative Treatment Of Intrabony Defect
- EPP Modified Technique+EMD+allograft+sCTG (Active Comparator): Procedure: After buccal intracervicular incision on vestibular aspects of two teeth surrounding the intrabony defect, a beveled vertical releasing incision was made in the buccal gingiva of the tooth affected by the intrabony defect, on the opposite site to the intrabony defect and extended beyond the mucogingival line to provide access to the intrabony defect. A buccal full thickness mucoperiosteal flap extending from the vertical incision to the defect-associated papilla and neigboring tooth was elevated. Interdental tunnel under the papillary tissue was elevated to the lingual bone crest. Granulation tissue and calculus from the inner aspect of papilla was removed.24%EDTA was applied on the exposed root surface, than rinsed and EMD and bone substitute was applied. sCTG taken form palate was sutured to the inner part of mucosa flap. Vertical incision was closed with simple single sutures, whereas due to modification of the original technique additional sling suture was applied.
  Interventions: Procedure: Modified Entire Papilla Preservation Technique (MEPPT) For Periodontal Regenerative Treatment Of Intrabony Defects.; Device: Emdogain (EMD), Biomaterials (allograft, subepithelial connective tissue graft/sCTG); Procedure: Modified Entire Papilla Preservation Technique (MEPPT) with Emdogain For Periodontal Regenerative Treatment Of Intrabony Defect; Procedure: Modified Entire Papilla Preservation Technique (MEPPT) with Emdogain and Allograft For Periodontal Regenerative Treatment Of Intrabony Defect; Procedure: Modified Entire Papilla Preservation Technique (MEPPT) with Emdogain and Allograft and sCTG For Periodontal Regenerative Treatment Of Intrabony Defect

INTERVENTIONS:
Procedure: Modified Entire Papilla Preservation Technique (MEPPT) For Periodontal Regenerative Treatment Of Intrabony Defects. — Surgical approach using modified papilla preservation technique for regenerative periodontal therapy.
Device: Emdogain (EMD), Biomaterials (allograft, subepithelial connective tissue graft/sCTG) — Surgical approach using modified papilla preservation technique and devices for regenerative periodontal therapy.
  Arms: EPP Modified Technique+EMD+allograft; EPP Modified Technique+EMD+allograft+sCTG; Entire Papilla Preservation Modified Technique + EMD
Procedure: Modified Entire Papilla Preservation Technique (MEPPT) with Emdogain For Periodontal Regenerative Treatment Of Intrabony Defect — Surgical approach using modified papilla preservation technique and Emdogain for regenerative periodontal therapy.
  Arms: EPP Modified Technique+EMD+allograft; EPP Modified Technique+EMD+allograft+sCTG; Entire Papilla Preservation Modified Technique + EMD
Procedure: Modified Entire Papilla Preservation Technique (MEPPT) with Emdogain and Allograft For Periodontal Regenerative Treatment Of Intrabony Defect — Surgical approach using modified papilla preservation technique and Emdogain and Allograft for regenerative periodontal therapy.
  Arms: EPP Modified Technique+EMD+allograft; EPP Modified Technique+EMD+allograft+sCTG
Procedure: Modified Entire Papilla Preservation Technique (MEPPT) with Emdogain and Allograft and sCTG For Periodontal Regenerative Treatment Of Intrabony Defect — Surgical approach using modified papilla preservation technique and Emdogain and Allograft and sCTG for regenerative periodontal therapy.
  Arms: EPP Modified Technique+EMD+allograft+sCTG

SUMMARY:
Regeneration of periodontal tissues is the primary goal of periodontal surgery regenerative procedures. Most techniques include an incision of the interdental papilla associated with defect. That may impair the volume and integrity of interdental tissues. Azzi et al. proposed a novel technique (Entire Papilla Preservation Technique, EPPT) for bone regeneration to secure the integrity of interdental papillae.

This study will search for differences in regeneration therapy of isolated interdental intrabony between Modified Entire Papilla Preservation Technique (MEPPT) alone and combined with EMD, demineralised freeze- dried bone allograft and sCTG. Moreover the aim of this study was to evaluate the clinical applicability and one- year outcomes in the regenerative treatment of isolated deep intrabony defects.

DETAILED DESCRIPTION:
Regeneration of periodontal tissues is the primary goal of periodontal surgery regenerative procedures. Both resorbable and nonresorbable barrier membranes have been widely used to receive periodontal regeneration, as well as different types of biomaterial have been investigated. Enamel matrix derivative (EMD, Emdogain, Straumann) become popular for periodontal regeneration, especially that membrane exposure due to bacterial contamination may deteriorate periodontal regeneration and wound healing especially in the interproximal areas. Hence different surgical procedures have been proposed to preserve interdental papilla. Most techniques include an incision of the interdental papilla associated with defect. That may impair the volume and integrity of interdental tissues. Azzi et al. proposed a novel technique (Entire Papilla Preservation Technique, EPPT) for bone regeneration to secure the integrity of interdental papillae by providing a tunnel- like undermining incision.

The completely preserved papillae improve wound healing process, stabilize the blood clot and the volume of interdental tissue. EMD and bone substitutes (allograft) are applied in the defect to promote periodontal regeneration. By using subepithelial connective tissue graft (sCTG) better quality (thickness) of soft tissue can be achieved. This clinical report describes surgical approach using modified papilla preservation technique for regenerative periodontal therapy. This study will search for differences in regeneration therapy of isolated interdental intrabony between Modified Entire Papilla Preservation Technique (MEPPT) alone and combined with EMD, demineralised freeze- dried bone allograft and sCTG. Moreover the aim of this study was to evaluate the clinical applicability and one- year outcomes in the regenerative treatment of isolated deep intrabony defects.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years (age 18-60 years), both genders
* Good compliance and good oral hygiene
* Systemically healthy
* Isolated intrabony defect of more than 3 mm depth, combined with more than 6 mm probing depth and attachment loss (stage III/IV periodontitis)
* The area of the intrabony defect should not exceed the lingual surface area of the root
* The morphology of the intrabony defect will be detected during the operation and finally determined whether the patient would be enrolled in the trial.
* The associated tooth should either maintain normal pulp vitality or should have undergone root canal therapy for at least 6 months before.

Exclusion Criteria:

* Full-mouth plaque index ≥ 20% (Ainamo & Bay 1975)
* Full-mouth sulcus bleeding index ≥ 15% (Mühlemann & Son 1971)
* Smoking
* Systemic diseases with compromised healing potential of infectious diseases
* Drugs affecting periodontal health / healing
* Pregnant and lactating females
* Previous periodontal surgery in the examined area
* Affected teeth with 3° mobility
* Furcation involvement
* Acute periapical inflammation

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 15 (Estimated)
Dates: Start 2021-09-10 (Actual); Primary Completion 2022-12-30 (Estimated); Study Completion 2023-09-01 (Estimated)

PRIMARY OUTCOMES:
Periodontal parameters measured before surgery. | 1-7 days before surgery
  1. Probing pocket depth (PPD) MEASURED IN MILIMETERS: distance from the gingival margin to the bottom of the gingival sulcus
  2. Clinical attachment level (CAL) MEASURED IN MILIMETERS: distance from the cementoenamel junction to the bottom of the gingival sulcus
  3. Recession height (RH) MEASURED IN MILIMETERS: distance from the cementoenamel junction to the gingival margin
  4. Width of keratinized tissue (WKT) MEASURED IN MILIMETERS: distance between the most apical point of the gingival margin and the mucogingival junction
  5. Gingival thickness (GT) MEASURED IN MILIMETERS: thickness of the gingiva measured 2-3 mm apical to the gingival margin
Periodontal parameters measured during surgery. | During surgery
  1. Intrabony component defects architecture after debridement MEASURED IN MILIMETERS(depth: distance between the crest of the marginal bone and the deepest location of the osseous defect, width: horizontal distance from the root surface to the alveolar bone crest).
  2. CEJ- BD, distance between cementoenamel junction and the bottom of the bone defect MEASURED IN MILIMETERS
Periodontal parameters measured on basis of X-ray | 1-7 days before surgery
  1. CEJ-MB: distance between cementoenamel junction (CEJ) and the crest of the marginal bone (MB) MEASURED IN MILIMETERS
  2. CEJ- BD: distance between cementoenamel junction (CEJ) and the bottom of the defect (BD) MEASURED IN MILIMETERS

SECONDARY OUTCOMES:
Periodontal parameters measured after surgery. | 12 months after surgery
  1. Probing pocket depth (PPD): distance from the gingival margin to the bottom of the gingival sulcus
  2. Clinical attachment level (CAL): distance from the cementoenamel junction to the bottom of the gingival sulcus
  3. Recession height (RH): distance from the cementoenamel junction to the gingival margin
  4. Width of keratinized tissue (WKT): distance between the most apical point of the gingival margin and the mucogingival junction
  5. Gingival thickness (GT): thickness of the gingiva measured 2-3 mm apical to the gingival margin
  6. Radiographic evaluation:
     1. Radiographical bone- filling of the intrabony defect
     2. CEJ- MB: distance between cementoenamel junction and the crest of the marginal bone
     3. CEJ- BD, distance between cementoenamel junction and the bottom of the bone defect
  ALL ABOVE PARAMETERS ARE MEASURED IN MILIMETERS

OTHER OUTCOMES:
Patient-reported outcomes based on VAS scales | 2 weeks after surgery
  Questionnaires:
  Scale 1: Pain after surgery (during recent 2 weeks) from 0 (no pain) to 10 (very big pain)
Patient-reported outcomes based on VAS scales | 2 weeks after surgery
  Scale 2: Eating disturbance (during recent 2 weeks) from 0 (no eating disturbance) to 10 (very big disturbance)
Patient-reported outcomes based on VAS scales | 2 weeks after surgery
  Scale 3: Daily functioning disturbance (during recent 2 weeks) from 0 (no daily functioning disturbance) to 10 (very big daily functioning disturbance)

CONTACTS AND LOCATIONS:
Overall Officials: Renata Górska, Professor, Study Chair — Department of Periodontal and Oral Mucosa Diseases in Warsaw
Locations (1):
- Department of Periodontology and Oral Mucosa Diseases, Medical University of Warsaw, Warsaw, Mazowsze, Poland

REFERENCES:
- [Derived] Gorski B, Jakubowska S, Wyrebek B. Entire Papilla Preservation Technique with Enamel Matrix Proteins and Allogenic Bone Substitutes for the Treatment of Isolated Intrabony Defects: A 3-Year Follow-Up of a Prospective Case Series. J Clin Med. 2025 Mar 30;14(7):2374. doi: 10.3390/jcm14072374. PMID 40217825